CLINICAL TRIAL: NCT01782027
Title: A Validation Study Evaluating the Use of 3H-Cholesterol Bound to Albumin as a Method to Assess Reverse Cholesterol Transport in Subjects With Monogenic Diseases Affecting HDL Metabolism
Brief Title: Mendelian Reverse Cholesterol Transport Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 815075
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cholesterol, HDL; Lipid Metabolism, Inborn Errors; Tangier Disease; LCAT Deficiency; Cholesteryl Ester Transfer Protein (CETP) Deficiency
Keywords: healthy controls; Tangier Disease; Adenosine triphosphate-binding cassette transporter 1 (ABCA1); apoA-I; LCAT deficiency; Scavenger receptor BI (SRBI) deficiency; CETP deficiency
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Tangier Disease; Lecithin Cholesterol Acyltransferase Deficiency; Cholesteryl Ester Transfer Protein Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3H-cholesterol (Experimental)
  Interventions: Drug: 3H-cholesterol bound to albumin

INTERVENTIONS:
Drug: 3H-cholesterol bound to albumin — up to 100 uCi of [3H]-cholesterol (containing approximately 0.2 mg of cholesterol) mixed with a solution containing human serum albumin will be administered as an intravenous bolus injection
  Other Names: particulate cholesterol

SUMMARY:
The purpose of this study is to investigate the use of radiolabeled particulate cholesterol administered intravenously in association with albumin, as a method to study reverse cholesterol transport (RCT) in people carrying mutations in genes known to affect high density lipoprotein (HDL) metabolism by analyzing changes in the tracer activity in total plasma, lipoproteins fractions and feces.

DETAILED DESCRIPTION:
The study will use 3H-cholesterol bound to albumin (particulate cholesterol) to assess the ability of HDL to transport cholesterol from the periphery to the liver to be eliminated. This process is called reverse cholesterol transport (RCT) and is one of the main mechanisms by which HDL protect against atherosclerotic cardiovascular disease. Mutations in some of the genes affecting HDL metabolism, may results in changes in RCT. The validation of a method assessing RCT is important for the development of new drugs which affect RCT and may result in useful treatments for atherosclerosis.

Subjects carrying mutations in genes known to affect HDL metabolism and healthy controls will be enrolled in the study. Changes in the tracer activity in total plasma, lipoproteins fractions and feces will be analyzed following the intravenous administration of radiolabeled particulate cholesterol.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 75
2. Subjects must be:

   1. Carriers of functional mutations of genes encoding proteins affecting HDL metabolism;
   2. Healthy control subjects with HDL cholesterol levels within the normal range of the lab where screening tests are run, or at the discretion of the investigator, and matched for gender, race, age (± 5 years) to the patients.
3. Negative screening pregnancy test if female of child bearing potential (females of child-bearing potential must be following a medically accepted form of contraception)
4. Subjects must be able to comprehend and willing to provide a signed IRB approved Informed Consent Form.
5. Subjects must be willing and able to comply with all study-related procedures.

Exclusion Criteria:

1. Known cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease (control subjects only)
2. History of diabetes mellitus or fasting glucose > 126 mg/dL at the screening visit (control subjects only).
3. Any current, unstable endocrine disease as assessed by collection of medical history during screening. Subjects with rare Mendelian disorders with thyroid disease that is well controlled by stable treatment may be considered for enrollment at the discretion of the principal investigator
4. History of previous malignancy, other than basal cell or squamous cell carcinoma of the skin, from which the patient has been disease free for less than 5 years as assessed by collection of medical history during screening
5. Current diagnosis of anemia as assessed by collection of medical history during screening or hemoglobin less than 10 g/dL as evaluated during safety lab at screening
6. History of kidney disease or chronic renal insufficiency, as defined as estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2 in control subjects and patients with other disorders of HDL metabolism and eGFR < 30 ml/min/1.73m2 in subjects with Lecithin-Cholesterol Acyltransferase (LCAT) deficiency.
7. Any active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition as assessed by collection of medical history during screening, and judged by the investigator to be a major condition.
8. Sustained uncontrolled hypertension (Systolic >160 mm Hg and/or Diastolic BP >100 mmHg) at screening. Blood pressure may be re-tested twice after initial assessment in the supine position at five minute intervals (for a total of 3 blood pressure assessments). The pressure elevation is considered sustained if either the systolic or the diastolic pressure values are outside the stated limits for all three assessments
9. Use of warfarin, or any known coagulopathy and /or elevated prothrombin time/partial thromboplastin time (PT/PTT) >1.5 x upper limit of normal (ULN)
10. Self-reported history of human immunodeficiency virus (HIV) positive
11. History of previous organ transplantation, as assessed by collection of medical history during screening
12. Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests such as alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5x ULN, or self-reported history of positive Hepatitis B or Hepatitis C test result
13. Any surgical procedure that occurred within the previous 3 months of the screening visit, as assessed by collection of medical history during screening, and judged by the investigator to be a major procedure.
14. History of drug abuse (< 1 year), as assessed by collection of medical history during screening procedures
15. Regular abuse of alcoholic beverages (> 2 drinks/day), as assessed by collection of medical history during screening procedures
16. Self-reported participation in an investigational drug study within 6 weeks prior to the screening visit
17. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study will be excluded.
18. Use of lipid lowering drugs expected to affect RCT (e.g. fibrates) within the 6 weeks prior to dosing or during the study, as assessed by collection of medical history during screening and concomitant medication checks at each study visit. Use of statins (stable dose for at least 30 days) is permitted.
19. Male subjects who plan to conceive a child within 3 months of the conclusion of the study.
20. Women who are pregnant or lactating or who are planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-10; Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
determination of 3H cholesterol in plasma and lipoproteins | up to 192 hr

SECONDARY OUTCOMES:
determination of 3H cholesterol and its metabolites in red blood cells over time | up to 192 hr

OTHER OUTCOMES:
determination of 3H cholesterol activity in feces | up to 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States